CLINICAL TRIAL: NCT04433013
Title: A Randomized Controlled Trial Assessing the Efficacy of Lianhua Qingwen as an Adjuvant Treatment in Patients With Mild Symptoms of COVID-19
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to find suitable site Principal Investigator. This study did not start and was withdrawn as of Aug 2020 (have updated as of Sept 2020, please proceed to update the status of study withdrawal accordingly)
Sponsor: Nanyang Technological University (Other)
Collaborators: Ministry of Health, Singapore (Other Government)
Responsible Party: Principal Investigator, Zhao Yan, Principal Investigator, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-2020-05-029
Record Dates: First submitted 2020-06-14; First posted 2020-06-16 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
Keywords: COVID-19; Traditional Chinese Medicine; Randomized Controlled Trial; Lianhua Qingwen
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Drug: Lianhua Qingwen
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lianhua Qingwen — The LHQW capsules will be administered to trial participants 4 capsules, 3 times a day, after meal
  Arms: Treatment group
Drug: Placebo — The placebo capsules will be administered to trial participants 4 capsules, 3 times a day, after meal
  Arms: Control group

SUMMARY:
COVID-19 virus remains in infected patients for extended periods of time. A great resource burden is placed on the healthcare system and society at large to isolate COVID-19 patients for prolonged periods. Thus, being able to increase the rate of viral clearance, thus reducing the duration of COVID-19 infection, would allow patients to be discharged earlier to free up resources for those who require it. The investigators designed a randomized controlled trial, investigating the use of Lianhua Qingwen, a TCM treatment, in COVID-19 infected patients with mild symptoms. The investigators hypothesize that the use of Lianhua Qingwen will increase the proportion of patients who test negative for COVID-19 after 8 days of TCM treatment when compared to the group of patients provided with standard care and placebo. Patients will be recruited from community isolation facilities, and have onset of symptoms within 5 days prior to admission to the isolation facility. The trial also evaluates the time taken for relief of clinical symptoms associated with COVID-19 and assesses the safety of the TCM treatment given to patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥21 years
2. Positive laboratory test for COVID-19 by RT-PCR methods
3. Presenting with at least one symptom (symptoms include fever, dry cough, sore throat, nasal congestion, malaise, headache, muscle pain, anosmia, and diarrhoea)
4. Length of time between date of onset of symptoms and the date of recruitment should not exceed 5 days to ensure that trial participants are in the early stages of infection
5. No clinical or radiographic evidence of pneumonia
6. Able to provide informed consent

Exclusion Criteria:

1. Individuals with underlying primary diseases such as cardiovascular, respiratory, liver, renal, diabetes, hepatitis A/B/C, gout or endocrinological diseases and neurological disorders which put them at a higher risk of developing severe disease
2. Individuals with compromised immune systems such as malignant tumors, organ or bone marrow transplants, HIV, or have taken immunosuppressants in the past three months.
3. Women who are pregnant or on lactation.
4. Individuals with mental illness.
5. History of allergy to any drug or food, or herb ingredient observed in this trial.
6. Individuals who are deemed not able to comply with trial procedure or follow-up

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who test negative for COVID-19 | after 8 days of treatment

SECONDARY OUTCOMES:
Time taken in days for relief of clinical symptoms | during the 8-day course of treatment
Proportion of participants with mild symptoms of COVID-19 progressing to moderate or severe illness | after 8 days of treatment and at the end of the trial
Proportion of participants who test positive for COVID-19 with Ct value>30 | after 8 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhao, Principal Investigator — Nanyang Technological University

IPD SHARING:
Plan to Share IPD: No